CLINICAL TRIAL: NCT02387749
Title: Effect Of Mesenchymal Stem Cells Transfusion on the Peripheral Neuropathy in Diabetic Patients Measured by Nerve Conduction.
Brief Title: Effect Of Mesenchymal Stem Cells Transfusion on the Diabetic Peripheral Neuropathy Patients .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, dina mohammed riad, Assistant Lecturer of Internal Medicine,faculty of medicine,Kasr Al Ainy hospital, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FACULTY OF MEDICINE,CAIRO U
Record Dates: First submitted 2015-03-01; First posted 2015-03-13 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetic peripheral neuropathy; mesenchymal stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cells (Experimental): The BM aspirate will be diluted at 6:1 ratio with phosphate buffer saline with 2 ml EDTA (30 ml BM aspirate+ 5 ml PBS/EDTA buffer).MNCs will be separated under aseptic conditions using a Ficoll. Hypaque desity gradient by centrifugation at 1800 rpm for 20 min then the MNCs will be plated in 40 ml(αMEM), serum free media; mesencult(MSCs culture),penicillin (100 U/ml),streptomycin(10 mg/ml),0.5 ml amphotericin B(all from Gibco BRL) and 10 ng/ml basic fibroblast growth factor (b-FGF)(R&D system, Minneapolis, MN) and will be incubated at 370 c in a humidified atmosphere containing 5% CO2 .after one day ,nonadherent cells will be cultured in the presence of Mesenchymal media for 3 weeks changed every week. After reaching 80% confluence the MSCs will be placed in 10 ml saline and infused IV.
  Interventions: Genetic: mesenchymal stem cells

INTERVENTIONS:
Genetic: mesenchymal stem cells — collection of stem cells by bone marrow biopsy from iliac crest, then culture for 1 month , then IV transfusion on 2 sessions to the same patient

SUMMARY:
A debilitating consequence of diabetes mellitus (DM) is neuropathy which globally affects between 20 -30% of diabetic patients and up to 50% in other studies. The incidence of diabetic neuropathy (DN) is estimated to be up to 45% for type 2 diabetic patients and 59% for type 1diabetic patients in USA.(DN) is the most common complication of DM.The pathophysiology of DN is promoted by several risk factors: micro vascular disease, neural hypoxia, and hyperglycemia-induced effects.At the molecular level, the primary cause of diabetic complications is known to be hyperglycemia, which disrupts cellular metabolism by the formation of reactive oxygen species (ROS).In the aspect of nerve functions, ROS formation increases neuron's susceptibility to damage. In addition, hyperglycemia impedes production of angiogenic and neurotrophic growth factors, which are necessary for normal function of neurons and glial cells and maintenance of vascular structure.No definitive disease-modifying treatments have been to reverse DN. The current treatment focuses on tight glycemic control which can reduce potential risk factors for further nerve damage and DN-associated pain management.In many studies, deficiency of neurotrophic factors and lack of vascular support have been regarded as key factors in the development DN.Mesenchymal stem cells (MSCs) are particularly attractive therapeutic agents because of their ability to self-renew, differentiate into multi lineage cell types, and locally secrete angiogenic cytokines, including basic fibroblast growth factor (bFGF) and vascular endothelial growth factor (VEGF) .These factors were reported to prompt neovascularization and have support for neural regeneration.It was plausible that MSCs may also be an effective therapeutic agent for the DN treatment through the paracrine effects of bFGF (Shibata et al., 2008) and VEGF and their potential to differentiate into neural cells such as astrocytes, oligodendrocytes , and Schwann cells.The adherent nature of MSCs makes them easy to expand in culture and an attractive candidate to use in cell therapy.Therefore, cell therapy has recently emerged as an attractive therapeutic strategy to meet the needs of both neurotrophic and vascular deficiencies of DN.Proper diagnosis of DN depends on the pattern of sensory loss, reflex test, electrodiagnostic studies, and imaging

DETAILED DESCRIPTION:
Objectives This study will be conducted to investigate the effects of Mesenchymal stem cells (MSC) transfusion on diabetic peripheral neuropathy in diabetic patient. (MSCs) have been reported to secrete various cytokines that exhibit angiogenic and neuro supportive effects.

Study Design Experimental interventional study. phase II clinical trial

Ethical committee approval (was it ethically approved by the department) Internal medicine department Yes

Study Methods

Population of study & disease condition (e.g women with hepatitis, ………) Diabetic patients(type I, type II) with documented peripheral neuropathy as determined by impaired nerve conduction

Inclusion criteria:

(Type I, type II) diabetic patients age range (18-45) years, with diabetic peripheral neuropathy proved by clinical assessment and nerve conduction who did not receive treatment for diabetic peripheral neuropathy.

Exclusion criteria:

Decompensated cardiac, renal or liver disease. Associated autoimmune diseases Associated endocrinal diseases Pregnancy, usage of contraceptive pills or steroids.

Methodology in details The study will be conducted on patients with diabetic peripheral neuropathy collected from internal medicine department(inpatient and out patients, males and females)

All subjects of this study will be submitted to the following :( preparatory visit before (MSCs) transfusion visit.)

* Thorough clinical assessment as a general assessment of the patient, also assessment of diabetes complications especially diabetic neuropathy. This is including full history and examinations (e.g., pain, sensory loss, ulcers, sensory level, etc….) this preparatory assessment will be done at internal medicine department.
* Venous blood will be drawn in the morning after an overnight fast in the pre (MSCs) transfusion visit.

Plasma biochemical blood measurements will be determined by standard laboratory procedures in the central lab at clinical pathology department, Kasr Alaini hospital)

* Fasting blood glucose level, 2 hours postprandial.
* C-peptide.
* Hb A1C.
* Basic Fibroblast Growth Factor (bFGF), vascular endothelial growth factor (VEGF) by ELISA.
* Complete blood picture.
* Liver functions in the form of ALT, AST
* Kidney functions in the form of serum creatinine.

  * fundus examination
  * Nerve conduction study at neurophysiology unit.
  * Bone marrow aspiration of about 90 ml under local anesthesia once at the first visit after preparatory visit mentioned before, the patient will be admitted for 12 hours and will be monitored closely to avoid anaphylaxis (by steroids, anti-allergic treatment), if no complication, will be discharged.

To avoid infection: During bone marrow aspiration, procedure will be done under complete aseptic precautions, placed in sterile tubes containing pre-servative-free heparin (Sigma-Aldrich, St. Louis, USA) Separation and processing of the sample will be done under good manufacture procedure (GMP): Bone Marrow Aspirate (BMA) will be withdrawn under good sterilization of the skin in an isolated area. Processing of the sample will be done in the laminar air flow; all supplies are disposable and sterile.

Technique:

Separation of mononuclear cells:

The bone marrow aspirate will be diluted at a ratio of 6:1 with phosphate buffer saline (PBS) with 2 mM EDTA (30 ml BM aspirate+ 5 ml PBS/EDTA buffer). The MNCs will be separated under aseptic conditions using a Ficoll. Hypaque desity gradient (density 1.077, GibcoBRL, Grand Islan, NY, USA) by centrifugation at 1800 rpm for 20 min then the MNCs will be plated in 40 ml alpha-modi-field Eagle's medium (αMEM), serum free media; mesencult(Mesenchymal stem cell culture),penicillin (100 U/ml),streptomycin(10 mg/ml),0.5 ml amphotericin B(all from Gibco BRL) and 10 ng/ml basic fibroblast growth factor (b-FGF) (R&D system, Minneapolis, MN) and will be incubated at 370 c in a humidified atmosphere containing 5% CO2 (Digirolamo et al.1999).after one day ,non adherent cells will be cultured in the presence of Mesenchymal media for 3 weeks changed every 1 week (cambrex Bioscience ,Nottingham, uk). After reaching 80% confluence the MSCs will be placed in 10 ml saline and will be infused intravenously

Flow cytometry Surface expression of MSCs using anti- (CD271, CD34, CD73, CD90, CD105, CD29) monoclonal antibodies (mAbs) will be analyzed using flow cytometry. MSCs (2X105 cells) will be suspended in PBS containing 1% BSA and will be stained with flurochrome -conjugated mAbs for 20 minutes on ice (anti-mouse mAanti-CD 271, CD34 CD73, CD90, CD105,CD29; BD Bioscience, MN, USA).flow cytometric analysis will be performed using a FACSCaliber (BD bioscience)equipped with cell Quest software.10000 cells will be passed in front of the laser for each sample. Each sample will be analyzed in duplicate. A cut off value at 20% will be set to categorize samples as positive.

Mesenchymal stem cells will be identified by morphology and immunophenotyping in the central lab at clinical pathology department, Kasr Alaini hospital( stem cell lab).

Mesenchymal stem cells transfusion slowly intravenous will be applied after these procedures for the patients after taking their approval and informed consent.

Follow up 3 months after Mesenchymal stem cells transfusion by fasting blood glucose level, 2 hours postprandial, C-peptide, Hb A1C, (bFGF), (VEGF) and nerve conduction at kasr Alaini hospital departments as mentioned before.

Possible Risk (mention if there is any risk or not) Anaphylaxis Infection

Primary outcomes (Most important outcomes to be assessed)

1- Effect of mesenchymal stem cells transfusion on diabetic peripheral neuropathy regarding improvement of clinical symptoms like pain, sensory loss and improvement of nerve conduction.

Secondary outcome parameters (other outcomes to be assessed)

1. Mesenchymal stem cells being a treatment modality in diabetes complications like peripheral neuropathy, to avoid hazards on patients secondary to diabetic peripheral neuropathy.
2. Improving of diabetic condition like lowering of blood glucose level, decrease in insulin requirements and improvement of general condition.

Sample size (number of participants included) 10 diabetic patients with diabetic peripheral neuropathy .

Source of funding (is there any source of funds or not) Faculty Of Medicine, Cairo University.

Time plan (when to start/ when expected to finish/ when to publish) At least 20 months

ELIGIBILITY:
Inclusion Criteria:

* (Type I, type II) diabetic patients age range (18-45) years, with diabetic peripheral neuropathy proved by clinical assessment and nerve conduction who did not receive treatment for diabetic peripheral neuropathy.

Exclusion Criteria:

* Decompensated cardiac, renal or liver disease. Associated autoimmune diseases Associated endocrinal diseases Pregnancy, usage of contraceptive pills or steroids.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gamal ElDin Saadi, phd, Study Chair — Cairo University; Dina Abdelmagid, MD, MRCP UK, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jackson L, Jones DR, Scotting P, Sottile V. Adult mesenchymal stem cells: differentiation potential and therapeutic applications. J Postgrad Med. 2007 Apr-Jun;53(2):121-7. doi: 10.4103/0022-3859.32215. PMID 17495381
- [Background] Keilhoff G, Stang F, Goihl A, Wolf G, Fansa H. Transdifferentiated mesenchymal stem cells as alternative therapy in supporting nerve regeneration and myelination. Cell Mol Neurobiol. 2006 Oct-Nov;26(7-8):1235-52. doi: 10.1007/s10571-006-9029-9. Epub 2006 Jun 16. PMID 16779672
- [Background] Kinnaird T, Stabile E, Burnett MS, Epstein SE. Bone-marrow-derived cells for enhancing collateral development: mechanisms, animal data, and initial clinical experiences. Circ Res. 2004 Aug 20;95(4):354-63. doi: 10.1161/01.RES.0000137878.26174.66. PMID 15321945
- [Background] Morbach S, Lutale JK, Viswanathan V, Mollenberg J, Ochs HR, Rajashekar S, Ramachandran A, Abbas ZG. Regional differences in risk factors and clinical presentation of diabetic foot lesions. Diabet Med. 2004 Jan;21(1):91-5. doi: 10.1046/j.1464-5491.2003.01069.x. PMID 14706061
- [Background] Nakae M, Kamiya H, Naruse K, Horio N, Ito Y, Mizubayashi R, Hamada Y, Nakashima E, Akiyama N, Kobayashi Y, Watarai A, Kimura N, Horiguchi M, Tabata Y, Oiso Y, Nakamura J. Effects of basic fibroblast growth factor on experimental diabetic neuropathy in rats. Diabetes. 2006 May;55(5):1470-7. doi: 10.2337/db05-1160. PMID 16644707
- [Background] Rathur HM, Boulton AJ. Recent advances in the diagnosis and management of diabetic neuropathy. J Bone Joint Surg Br. 2005 Dec;87(12):1605-10. doi: 10.1302/0301-620X.87B12.16710. No abstract available. PMID 16326870
- [Background] Shibata T, Naruse K, Kamiya H, Kozakae M, Kondo M, Yasuda Y, Nakamura N, Ota K, Tosaki T, Matsuki T, Nakashima E, Hamada Y, Oiso Y, Nakamura J. Transplantation of bone marrow-derived mesenchymal stem cells improves diabetic polyneuropathy in rats. Diabetes. 2008 Nov;57(11):3099-107. doi: 10.2337/db08-0031. Epub 2008 Aug 26. PMID 18728233
- [Background] Adler AI, Stratton IM, Neil HA, Yudkin JS, Matthews DR, Cull CA, Wright AD, Turner RC, Holman RR. Association of systolic blood pressure with macrovascular and microvascular complications of type 2 diabetes (UKPDS 36): prospective observational study. BMJ. 2000 Aug 12;321(7258):412-9. doi: 10.1136/bmj.321.7258.412. PMID 10938049
- [Background] Digirolamo CM, Stokes D, Colter D, Phinney DG, Class R, Prockop DJ. Propagation and senescence of human marrow stromal cells in culture: a simple colony-forming assay identifies samples with the greatest potential to propagate and differentiate. Br J Haematol. 1999 Nov;107(2):275-81. doi: 10.1046/j.1365-2141.1999.01715.x. PMID 10583212
- [Background] Dalla Paola L, Faglia E. Treatment of diabetic foot ulcer: an overview strategies for clinical approach. Curr Diabetes Rev. 2006 Nov;2(4):431-47. doi: 10.2174/1573399810602040431. PMID 18220646
- [Derived] Aldali F, Deng C, Nie M, Chen H. Advances in therapies using mesenchymal stem cells and their exosomes for treatment of peripheral nerve injury: state of the art and future perspectives. Neural Regen Res. 2025 Nov 1;20(11):3151-3171. doi: 10.4103/NRR.NRR-D-24-00235. Epub 2024 Oct 22. PMID 39435603

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesenchymal Stem Cells Transfusion in Diabetic Neuropathy: collection: bone marrow biopsy from iliac crest. Separation of cells:The bone marrow aspirate will be diluted at a ratio of 6:1 with phosphate buffer saline (PBS) with 2 ml EDTA (30 ml BM aspirate+ 5 ml PBS/EDTA buffer). The MNCs will be separated under aseptic conditions using a Ficoll. Hypaque desity gradient by centrifugation at 1800 rpm for 20 min then the MNCs will be plated in 40 ml alpha-modi-field Eagle's medium (αMEM), serum free media; mesencult(Mesenchymal stem cell culture),penicillin (100 U/ml),streptomycin(10 mg/ml),0.5 ml amphotericin B(all from Gibco BRL) and 10 ng/ml basic fibroblast growth factor (b-FGF) (R&D system, Minneapolis, MN) and will be incubated at 37 c in a humidified atmosphere containing 5% CO2.after one day,non adherent cells will be cultured in the presence of Mesenchymal media for 3 weeks changed every 1 week. After reaching 80% confluence the MSCs will be placed in 10 ml saline and will be infused intravenously. on 2 sessions to the same patient
Period: Overall Study
Arm/Group | Mesenchymal Stem Cells Transfusion in Diabetic Neuropathy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: blood pressure all patients were normal blood pressure measurement
  routine lab investigations were normal to exclude other co-morbidites
Groups:
- Mesenchymal Stem Cells Transfusion in DPN Patients: This study was conducted on 10 patients with Diabetic peripheral neuropathy (DPN), 4 females and 6 males
Arm/Group | Mesenchymal Stem Cells Transfusion in DPN Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.20 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Egypt | 10

OUTCOME MEASURES:

1. Primary Outcome: Measurement of b-FGF, v-EGF MEASURED BY ELISA
Description: measurement of b-FGF and v-EGF MEASURED BY ELISA before (at zero), and after at (7 days, 90) days after stem cell transfusion to measure the effect of stem cell and its role in nerve regeneration
Time Frame: zero ( before) , 7 DAYS, 90 days
Population: b-FGF, V-EGF (pg/ml) measured at zero, 7 days after stem cell transfusion measured by ELISA to measure the effectiveness of stem cells and as an indication for nerve regeneration
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Measurement of b-FGF and v- EGF MEASURED BY ELISA: measurement of b-FGF and v- EGF MEASURED BY ELISA before (at zero), and after at (7 days, 90) days after stem cell transfusion to measure the effect of stem cell and its role in nerve regeneration
Arm/Group | Measurement of b-FGF and v- EGF MEASURED BY ELISA
Number analyzed (Participants) | 10
pg/ml
  b-FGF ZERO | 30.2 (16.7)
  b-FGF 7 DAYS | 55.4 (12.3)
  b-FGF 90 days | 30.3 (14.8)
  v- EGF ZERO | 428.7 (125)
  v- EGF 7 DAYS | 601.8 (141.8)
  v-EGF 90 DAYS | 371.5 (121.9)
Statistical Analysis 1: Comparison: Measurement of b-FGF and v- EGF MEASURED BY ELISA; Test type: Superiority; p = 0.005, Chi-squared, Corrected

2. Primary Outcome: Change of Nerve Conduction Velocities of Nerves Affected Measured by Nerve Conduction Study.
Description: Measuring nerve conduction velocities(NCV) in m/sec upper and lower limbs nerves(sensory and motor) lower limb nerves : tibial , common peroneal(CP) as motor and sural nerve as sensory upper limb nerves: ulnar nerve as motor and sensory and compare at base line(zero day) and 90 days after stem cells transfusion
Time Frame: base line(zero dya), 90 days after stem cells transfusion.
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- Nerve Conduction Velocities of Nerves: nerve conduction velocities of nerves examined measured in Upper limbs and Lower limbs nerves,motor and sensory
  lower limb motor nerves: tibial and common peroneal lower limb sensory nerve : sural nerve
  upper limb motor nerve: ulnar nerve upper limb sensory nerve: ulnar nerve
  data measured at zero (before stem cell transfusion) and 90 days after stem cell transfusion
Arm/Group | Nerve Conduction Velocities of Nerves
Number analyzed (Participants) | 10
m/sec
  Tibial Motor Nerve conduction velocity zero | 43.6 (8.5)
  Tibial motor nerve conduction velocity 90 days | 44.4 (6.6)
  common peroneal motor nerve velocity at zero day | 43.8 (10.3)
  common peroneal motor nerve velocity at 90 day | 45.2 (12.3)
  Ulnar Motor Nerve conduction velocity at zero day | 56.0 (8.7)
  Ulnar Motor Nerve conduction velocity at 90 days | 54.2 (10.6)
  Ulnar sensory Nerve conduction velocity zero day | 52.0 (16.3)
  Ulnar sensory Nerve conduction velocity at 90 days | 51.2 (12.4)
  Sural Nerve conduction Velocity at zero day | 21.1 (22.7)
  Sural Nerve conduction Velocity at 90 days | 25.5 (27.0)

3. Primary Outcome: Change of Nerve Conduction Latency of Nerves Affected Measured by Nerve Conduction Study
Description: Measuring nerve conduction latency in msec of upper and lower limbs nerves(sensory and motor) lower limb nerves : tibial , common peroneal(CP) as motor and sural nerve as sensory upper limb nerves: ulnar nerve as motor and sensory and compare at base line and 90 days after stem cells transfusion
Time Frame: base line(zero dya), 90 days after stem cells transfusion .
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Nerve Conduction Latency of Nerves: nerve conduction latency of nerves examined measured in Upper limbs and Lower limbs nerves,motor and sensory lower limb motor nerves: tibial and common peroneal lower limb sensory nerve : sural nerve upper limb motor nerve: ulnar nerve upper limb sensory nerve: ulnar nerve data measured at zero (before stem cell transfusion) and 90 days after stem cell transfusion
Arm/Group | Nerve Conduction Latency of Nerves
Number analyzed (Participants) | 10
msec
  Tibial Motor nerve conduction latency zero day | 4.4 (1.9)
  Tibial Motor nerve conduction latency 90 days | 4.1 (1.3)
  common peroneal motor nerve latency at zero day | 4.4 (1.8)
  common peroneal motor nerve latency at 90 day | 4.2 (1.1)
  Ulnar Motor Nerve conduction latency at zero day | 2.9 (0.8)
  Ulnar Motor Nerve conduction latency at 90 day | 2.9 (0.7)
  Ulnar sensory Nerve conduction latency zero day | 3.0 (1.0)
  Ulnar sensory Nerve conduction latency 90 days | 2.7 (0.8)
  Sural Nerve conduction latency at zero day | 2.2 (2.4)
  Sural Nerve conduction latency at 90 days | 2.5 (2.8)

4. Primary Outcome: Change of Nerve Conduction Amplitude of Nerves Affected Measured by Nerve Conduction Study.
Description: Measuring nerve conduction amplitudes in uv of upper and lower limbs nerves(sensory and motor).
  lower limb nerves : tibial , common peroneal(CP) as motor and sural nerve as sensory .
  upper limb nerves: ulnar nerve as motor and sensory. and compare at base line and 90 days after stem cells transfusion
Time Frame: base line(zero dya), 90 days after stem cells transfusion
Measure: Mean (Standard Deviation); unit: uv
Groups:
- Nerve Conduction Amplitudes of Nerves: nerve conduction amplitudes of nerves examined measured in Upper limbs and Lower limbs nerves,motor and sensory lower limb motor nerves: tibial and common peroneal, lower limb sensory nerve : sural nerve.
  upper limb motor nerve: ulnar nerve motor , upper limb sensory nerve: ulnar nerve sensory data measured at zero (before stem cell transfusion) and 90 days after stem cell transfusion
Arm/Group | Nerve Conduction Amplitudes of Nerves
Number analyzed (Participants) | 10
uv
  Tibial Motor nerve Amplitude zero day | 3.8 (4.0)
  Tibial Motor nerve Amplitude at 90 days | 3.4 (3.0)
  common peroneal motor nerve amplitude at zero day | 2.2 (1.9)
  common peroneal motor nerve amplitude at 90 days | 2.2 (1.2)
  Ulnar Motor Nerve conduction amplitude zero day | 5.4 (1.9)
  Ulnar Motor Nerve conduction amplitude at 90 days | 6.3 (1.8)
  Ulnar sensory Nerve conduction amplitude zero day | 23.1 (16.5)
  Ulnar sensory Nerve conduction amplitude at 90 day | 21.3 (11.6)
  Sural Nerve conduction amplitude at zero day | 5.2 (5.8)
  Sural Nerve conduction amplitude at 90 day | 7.3 (8.6)

5. Secondary Outcome: Change of Levels of Fasting Blood Sugar and 2 Hours Post Prandial at Base Line ( Zero Day ) and After (90 Days) After Stem Cells Transfusion
Description: fasting, 2 hours postprandial blood sugar measurement before at base line (zero day) and after (90 days) stem cells transfusion as a follow up and comparing the values.
Time Frame: base line (zero day) and 90 days after stem cells transfusion
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Blood Tests Measured Before and After Stem Cell Transfusion: Plasma biochemical blood measurements will be determined by standard laboratory procedures in the central lab at clinical pathology department, Kasr Alaini hospital) Fasting blood glucose level, 2 hours postprandial.
Arm/Group | Blood Tests Measured Before and After Stem Cell Transfusion
Number analyzed (Participants) | 10
mg/dl
  fasting blood sugar zero | 211.30 (61.92)
  fasting blood sugar 90 days | 145.70 (37.56)
  2 hours post postprandial blood sugar Zero | 291.50 (106.56)
  2 hours post postprandial blood sugar 90 days | 190.30 (56.42)

6. Secondary Outcome: Change of Levels of Glycated Haemoglobin( HA1C) After Stem Cells Transfusion Measured in Percent %
Description: Blood tests before and after stem cells(90 days) transfusion and comparing the values in percent % which is reflecting the patient blood sugar control in the previous 3 months
Time Frame: at base line (zero day) and 90 days after stem cells transfusion
Measure: Mean (Standard Deviation); unit: percent %
Groups:
- HA1C Measurment Before and Afterr Stem Cell: as a cumulative effect of patient control we measured HA1C at zero level and 90 days after stem cell transfusion in %
Arm/Group | HA1C Measurment Before and Afterr Stem Cell
Number analyzed (Participants) | 10
percent %
  HA1C Level Zero | 9.12 (3.42)
  HA1C Level 90 days | 7.96 (1.89)

ADVERSE EVENTS:
Time Frame: 3 months
Description: monitoring to mainly anaphylaxis and risk of infection which are the main side effects after stem cells infusion were recorded and excluded.
  regular follow up monthly up to 3 months recorded without serious side effects.
Arm/Group | Mesenchymal Stem Cells Transfusion in Diabetic Neuropathy
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
patients are not so co-operative regarding stem cell collection by bone marrow biopsy, Lab requirements for stem cell culture and follow up are limited to the university lab with expensive equipment and kits The sample is small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes